CLINICAL TRIAL: NCT07221669
Title: An Open-Label Study to Assess the Efficacy and Safety of Multiple Doses of Salanersen (BIIB115) Delivered Intrathecally to Treatment-Naïve, Presymptomatic Infants With Genetically Diagnosed Spinal Muscular Atrophy
Brief Title: A Study to Learn About Salanersen's (BIIB115) Effects on Movement and Its Safety When Given Before Symptoms Appear in Babies With Genetically Diagnosed Spinal Muscular Atrophy (SMA)
Acronym: STELLAR-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 277SM302; 2025-523116-37 (Other: EU CTIS Number)
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Salanersen (Experimental): In Part 1 of the study, participants will receive two doses of salanersen, 80 milligrams (mg) by intrathecal (IT) lumbar puncture (LP), approximately 12 months apart. Participants who complete Part 1 of the study will receive three doses of salanersen, 80 mg by IT LP, approximately 12 months apart, in Part 2 of the study.
  Interventions: Drug: Salanersen

INTERVENTIONS:
Drug: Salanersen — Administered intrathecally
  Other Names: BIIB115

SUMMARY:
In this study, researchers will learn more about the effects and safety of BIIB115, also known as salanersen.

Specifically, researchers will learn more about how salanersen works in babies who have been diagnosed with SMA through genetic testing but have not yet started showing signs or symptoms. Most people with SMA have changes in a gene called survival motor neuron 1, also known as SMN1. These changes lower the amount of SMN protein in their bodies. Without enough of this protein, motor neurons and muscles cannot work properly. A similar gene called SMN2 can help replace some of the lost SMN protein in the body. Salanersen works by helping the SMN2 gene to make more SMN protein.

In this study, participants will have either 2 SMN2 copies or 3 SMN2 copies. The higher the copy number, the less severe the participant's SMA is.

The main goal of this study is to see if starting salanersen before signs or symptoms appear can prevent signs or symptoms of SMA or make them less severe. Researchers will use different tests to learn if motor symptoms are changing, including the World Health Organization (WHO) motor milestones.

The main questions researchers want to answer in this study are:

* How many participants with 2 copies of the SMN2 gene can sit without support at 12 months?
* How many participants with 3 copies of the SMN2 gene can walk alone at 18 months?

Researchers will also learn more about:

* The effects on participants' motor symptoms and how many new movement milestones participants achieve.
* How many participants stay free of SMA symptoms
* How much salanersen gets into the fluid surrounding the brain and spinal cord.
* How much salanersen gets into the blood.
* How many participants have adverse events or serious adverse events. Adverse events are health problems that may or may not be caused by the study drug.

This study will be done as follows:

* First, participants will be screened to check if they can join the study. The screening period will be up to 28 days.
* This is an "open label" study. This is a study in which the participants, study doctor, and site staff know which study drug participants are receiving. In this study, all participants will receive salanersen through an intrathecal injection, or one that is given into the fluid surrounding the brain and spinal cord.
* There will be 2 parts in this study. During Part 1, participants will receive 2 doses of salanersen, about 12 months apart from each other. Part 1 will last up to 25 months.
* During Part 2, participants will continue to receive salanersen. They will receive up to 3 doses, 12 months apart from each other. Part 2 will last up to 36 months.
* During Part 1, participants will have up to 11 clinic visits and up to 3 phone calls. During Part 2, participants will have up to 7 clinic visits and up to 12 phone calls.

DETAILED DESCRIPTION:
For Part 1 of the study, the primary objective is to evaluate the clinical efficacy of salanersen in participants with genetically diagnosed SMA, and the secondary objective is to evaluate safety and tolerability, pharmacokinetics (PK), and effect on biomarkers after treatment with salanersen in participants with genetically diagnosed SMA.

For Part 2 of the study, the primary objective is to evaluate the long-term clinical efficacy of salanersen in participants with genetically diagnosed SMA, and the secondary objective is to evaluate the long-term safety and tolerability, PK, and effect on biomarkers after treatment with salanersen in participants with genetically diagnosed SMA.

ELIGIBILITY:
Key Inclusion Criteria:

-≤42 days of age at first dose of salanersen.

* Genetic documentation of 5q SMA homozygous gene deletion or mutation or compound heterozygous mutation.
* Two or three copies of the survival motor neuron 2 (SMN2) gene.
* Ulnar compound muscle action potential (CMAP) amplitude ≥2 millivolt (mV) at Screening and Day 1 predose.
* Body weight ≥3rd percentile for age based on World Health Organization (WHO) Child Growth Standards at the time of informed consent.

Key Exclusion Criteria:

* Any clinical signs or symptoms at Screening or Day 1 predose that are, in the opinion of the Investigator, strongly suggestive of SMA.
* Areflexia on neurologic examination at biceps, knee, or ankle at Screening or Day 1 Predose.
* Hypoxemia (oxygen saturation <96% awake or asleep without any supplemental oxygen or respiratory support, or for altitudes >1000 meters (m), oxygen saturation of <92% awake or asleep without any supplemental oxygen or respiratory support).
* Diagnosis of neonatal respiratory distress syndrome necessitating surfactant replacement therapy or invasive ventilatory support.
* Any reason, anatomical or otherwise (including hematology/coagulation laboratory results), that presents increased risk of complication from the LP procedures or safety assessments.
* Any prior treatment with an approved SMA disease-modifying therapy (e.g., nusinersen, onasemnogene abeparvovec-xioi [OA], and/or risdiplam), a myostatin inhibitor therapy, or an investigational drug given for the treatment of SMA.

Note: Other protocol-defined inclusion/exclusion criteria will apply.

Ages: 0 Days to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-11-28 (Estimated); Study Completion 2032-05-29 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of Participants with 2 Survival Motor Neuron 2 (SMN2) Copies Sitting Without Support (for at Least 10 Seconds) | At Month 12
Part 1: Percentage of Participants with 3 SMN2 Copies Walking Alone (for at Least 5 Steps) | At Month 18
Part 2: Percentage of Participants Attaining and Maintaining World Health Organization (WHO) Motor Milestones | Up to Day 1825
  The WHO motor milestones will include six key developmental milestones: sitting without support, standing with assistance, hands-and-knees crawling, walking with assistance, standing alone, and walking alone.

SECONDARY OUTCOMES:
Part 1: Percentage of Participants Attaining World Health Organization (WHO) Motor Milestones | Up to Day 730
  The WHO motor milestones will include six key developmental milestones: sitting without support, standing with assistance, hands-and-knees crawling, walking with assistance, standing alone, and walking alone.
Parts 1 and 2: Percentage of Participants Attaining Hammersmith Infant Neurological Examination Section 2 (HINE-2) Motor Milestones | Up to Day 1825
  Section 2 of the HINE is used to assess motor milestones and includes 8 motor milestone categories: voluntary grasp (0 to 3), ability to kick in supine position (0 to 4), head control (0 to 2), rolling (0 to 3), sitting (0 to 4), crawling (0 to 4), standing (0 to 3), and walking (0 to 3). Total HINE-2 score is the sum of points from each item and can range from 0 to 26, with higher scores depicting a better level of ability.
Parts 1 and 2: Change From Baseline in Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) Motor Function Scale | Up to Day 1825
  The CHOP INTEND test is designed to evaluate the motor skills of participants with significant motor weakness. It includes 16 items (capturing neck, trunk, and proximal and distal limb strength) structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). All item scores range from 0-4. The total score ranges from 0-64, with higher scores depicting better motor function.
Parts 1 and 2: Change From Baseline in Compound Muscle Action Potential (CMAP) Amplitudes | Up to Day 1825
  CMAP is a well validated method for tracking disease progression in neuromuscular disorders such as SMA and amyotrophic lateral sclerosis and has been proposed as a potential biomarker of a therapeutic effect in SMA. CMAPs will be performed for the following nerve-muscle pairs: ulnar-abductor digiti minimi and peroneal-tibialis anterior.
Part 1: Percentage of Participants who Remain Free of Clinically Manifested Spinal Muscular Atrophy (SMA) | Up to Day 730
Part 2: Hammersmith Functional Motor Scale Expanded (HFMSE) Total Score | Up to Day 1825
  The HFMSE is a tool used to assess motor function in individuals with SMA. Participants will be asked to complete a specific movement and are then graded on the quality and execution of that movement. Higher scores indicate higher levels of motor ability. The overall score is the sum of the scores for all 33 items, with a maximum score of 66 with higher scores depicting better ability to perform activities.
Part 2: Change From Baseline in Hammersmith Functional Motor Scale Expanded (HFMSE) | Up to Day 1825
  The HFMSE is a tool used to assess motor function in individuals with SMA. Participants will be asked to complete a specific movement and are then graded on the quality and execution of that movement. Higher scores indicate higher levels of motor ability. The overall score is the sum of the scores for all 33 items, with a maximum score of 66 with higher scores depicting better ability to perform activities.
Part 2: Revised Upper Limb Module (RULM) Total Score | Up to Day 1825
  The RULM is developed to assess upper limb functional abilities of participants with SMA. This test consists of a total of 20 upper limb performance items that are reflective of activities of daily living. The RULM is scored from 0 to 37 points, with higher scores indicating better function.
Part 2: Change From Baseline in Revised Upper Limb Module (RULM) | Up to Day 1825
  The RULM is developed to assess upper limb functional abilities of participants with SMA. This test consists of a total of 20 upper limb performance items that are reflective of activities of daily living. The RULM is scored from 0 to 37 points, with higher scores indicating better function.
Part 2: Percentage of Participants who Develop Spinal Muscular Atrophy (SMA) Subtypes (Type 1, 2,3a and 3b) As Assessed by the Investigator | Up to Day 1825
Parts 1 and 2: Time to Death (Overall Survival) | Up to Day 1825
Parts 1 and 2: Time to Death or Permanent Ventilation | Up to Day 1825
  Permanent ventilation is defined as tracheostomy or ≥16 hours ventilation/day continuously for >21 days in the absence of an acute reversible event.
Parts 1 and 2: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 1825
Parts 1 and 2: Concentration of Salanersen in Cerebrospinal Fluid (CSF) | Up to Day 1460
Parts 1 and 2: Concentration of Salanersen in Serum | Up to Day 1825
Parts 1 and 2: Change From Baseline in Plasma Levels of Neurofilament Light Chain (NfL) | Up to Day 1825

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Neurology Rare Disease Center, Flower Mound, Texas
  - Childrens Hospital of the Kings Daughter Norfolk, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/